CLINICAL TRIAL: NCT06137807
Title: A Prospective, Multicenter Clinical Trial of the TricValve® Transcatheter Bicaval Valve System in Subjects With Severe Tricuspid Regurgitation - TRICAV-I Trial
Brief Title: TRIcvalve biCAVal Valve System for Severe Tricuspid Regurgitation (TRICAV-I)
Acronym: TRICAV-I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: P+F Products + Features USA Inc. (Industry)
Collaborators: P+F Products + Features GmbH (Industry); Meditrial USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-TRIC-005
Record Dates: First submitted 2023-10-31; First posted 2023-11-18 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Tricuspid Regurgitation; Tricuspid Valve Disease
Keywords: Tricuspid Regurgitation; Heart Failure
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Failure

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter clinical trial. Subjects will be selected by their local Heart Team to be at high risk and deemed eligible by an independent eligibility committee (IEC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- TricValve® Device (Device) Group (Experimental): subjects will undergo TricValve® implantation and will continue to be managed with optimal medical therapies, per physician discretion.
  Interventions: Device: TricValve® Transcatheter Bicaval Valve System

INTERVENTIONS:
Device: TricValve® Transcatheter Bicaval Valve System — The TricValve® Transcatheter Bicaval Valve System is a bicaval transcatheter tricuspid valve replacement system, which includes the TricValve® Transcatheter Bicaval Valve for superior vena cava (SVC) and the TricValve® Transcatheter Bicaval Valve for inferior vena cava (IVC). The system is a single use, sterile device compatible with all the valve sizes. The valves are premounted in the TricValve® Delivery System. The prostheses are implanted percutaneously into the inferior and superior vena cava without disturbing the native tricuspid valve. The device is made of bovine pericardium leaflets sutured on a nitinol self-expanding stent system available in sizes 25 and 29 for superior vena cava and 31 and 35 for inferior vena cava. The valve is implanted percutaneously by the transfemoral approach. The valves are supplied already premounted into the TricValve® Delivery System.
  Other Names: TricValve System

SUMMARY:
The TricValve® Transcatheter Bicaval Valve System is a bicaval transcatheter tricuspid valve replacement system, which includes the TricValve® Transcatheter Bicaval Valve for superior vena cava (SVC) and the TricValve® Transcatheter Bicaval Valve for inferior vena cava (IVC). The TricValve® Transcatheter Bicaval Valves are pre-mounted into the TricValve® Delivery System which is used for percutaneous access and delivery of the TricValve® Transcatheter Bicaval Valve in the vena cava. The system is a single use, sterile device compatible with all the valve sizes. The prostheses are implanted percutaneously into the inferior and superior vena cava without disturbing the native tricuspid valve. The device is made of bovine pericardium leaflets sutured on a nitinol self-expanding stent system.

DETAILED DESCRIPTION:
This is a prospective multicenter clinical investigation designed to evaluate the safety and effectiveness of the TricValve® Transcatheter Bicaval Valve System for improving outcomes in symptomatic subjects with severe TR deemed by the local Heart Team to be at high risk for tricuspid valve surgery.

Patients who meet all of the study inclusion criteria, will be treated with the TricValve System. After the intervention, patients will be followed up closely for 12 months. Long term safety and efficacy data will be collected annually up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 years or older, at the time of signing the informed consent.
2. Subjects has severe tricuspid regurgitation (TR), as determined by the qualifying transthoracic echocardiogram (TTE) confirmed by an echocardiography Core Lab.
3. NYHA Class III-IVa (not on inotropes, IABP or LVAD) or heart failure (HF) admission in the past 6 months.
4. Subject is adequately treated with optimal medical therapy (OMT) for heart failure per the local Heart Team for at least 30 days prior to the index procedure, including a diuretic.
5. The local Heart Team and IEC determine that the patient is eligible for the TricValve procedure.
6. For females of childbearing potential, negative pregnancy test.
7. Capable of giving signed informed consent.

Exclusion Criteria:

1. Subject had a recent MI, stroke or cardiovascular accident; underwent coronary artery bypass graft surgery, had a percutaneous coronary intervention or other major cardiovascular surgery within 90 days prior to TricValve implantation.
2. Subject requires another planned major cardiac procedure, including left-sided transcatheter intervention or surgery (e.g. severe aortic stenosis, severe mitral regurgitation), coronary artery bypass or PCI or pulmonary valve correction. Please note that if closure of an ASD, iatrogenic ASD or PFO is performed, TricValve implantation can be performed 30 days after the intervention. Additionally, TricValve implantation can be performed 30 days after any Electrophysiology procedure (pacemaker, ICD, etc.).
3. LVEF ≤ 30% on echocardiography.
4. Evidence of intracardiac, inferior vena cava (IVC), or femoral venous mass, thrombus or vegetation.
5. Tricuspid stenosis. (Per TVARC, echo criteria: TVA at least 1.5 cm2 or TVAi at least 0.9 cm2/m2 [at least 0.75 if BMI >30 kg/m2], DVI <2.2, mean gradient <5mm Hg); reduction of total tricuspid regurgitation to optimal (≤ mild [1+]) or acceptable (≤ moderate [2+]).
6. Severe right ventricular dysfunction.
7. Cardiac amyloidosis
8. Pulmonary artery systolic pressure (PASP) >65 mmHg assessed with Echo Doppler and /or right heart catheterization.
9. Lower extremity venous thrombosis and/or the presence of an IVC filter at the time of or 6 months prior to TricValve procedure.
10. Hemodynamically significant pericardial effusion.
11. Patient with refractory heart failure requiring advanced intervention (i.e. left ventricular assist device, transplantation) (ACC/ AHA/ ESC/ EACTS Stage D heart failure)
12. Any known allergy or hypersensitivity to nitinol, bovine tissue or contrast media that cannot be adequately treated with pre-medication.
13. Unable to tolerate anticoagulation/antiplatelet therapy
14. Hemodynamic instability, cardiogenic shock, inotropic support, intra-aortic balloon pump or acute heart failure within 30 days prior to the TricValve procedure.
15. Any known life-threatening condition with an estimated life span of at least 12 months.
16. Platelet count < 75,000/mm3
17. Child-Pugh Severity Class C (10-15 points).
18. Severe renal insufficiency with estimated glomerular filtration rate (eGFR) ≤ 25 mL/min/1.73 m2 or requiring chronic renal replacement therapy at the time of enrollment.
19. Endocarditis or active/ongoing infection requiring antibiotics.
20. Unable to walk at least 60 meters in a 6minute walk test.
21. Known bleeding or clotting disorders or patient refuses blood transfusion.
22. Active gastrointestinal (GI) bleeding within 3 months of randomization.
23. Presence of significant congenital heart disease including but not limited to hemodynamically significant atrial septal defect, RV dysplasia, and arrhythmogenic RV.
24. Use or participation in other investigational device or drug study in which patient has not reached a primary endpoint to treat cardiovascular conditions related to the outcomes of the current study.
25. Any other condition that would preclude ability to meet study requirements in the opinion of the investigator.
26. Psychiatric/behavioral issues or other medical or social conditions that preclude valid consent and follow-up
27. Pregnant or breastfeeding subjects and those who plan pregnancy during the clinical investigation follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 Month and 12 Months
  Number of days until death
Stroke | 1 Month
  Number of days until death
Pulmonary Embolism | 1 Month
  Number of days until death
Valve Academic Research Consortium (VARC) type 2-4 bleeding complication | 1 Month
  Number of days until death
Major vascular, access-related, or cardiac structural complication | 1 Month
  Number of days until death
Stage 3 Acute Kidney Injury with increase in serum creatinine >300% (>3.0x increase) and/or serum creatinine ≥4.0mg/dL (≥354 μmol/L) with an acute increase of ≥ 0.5 mg/dL (≥44 μmol/L) | 7 Days
  Number of days from baseline until increase
Stage 4 Acute Kidney Injury requiring new temporary or permanent renal replacement therapy | 1 Month
  Number of days until new renal replacement therapy
Emergency surgery or intervention related to the device/procedure complications | 1 Month
  Number of days until emergency surgery or intervention
Right Ventricular Assist Device (RVAD) implantation or heart transplant | 12 Months
  Number of days until Right Ventricular Assist Device (RVAD) implantation or heart transplant
Tricuspid valve surgery or percutaneous tricuspid intervention | 12 Months
  Number of days until tricuspid valve surgery or percutaneous tricuspid intervention
Heart Failure Events | 12 Months
  Number of heart failure episodes including hospitalization, or worsening heart failure
Kansas City Cardiomyopathy Questionnaire (KCCQ) Score | 12 Months
  Change in KCC score (score ranges between 0 and 100)
New York Heart Association (NYHA class) | 12 Months
  Change in NYHA class (range from I to IV)
Six Minute Walking Test (6MWT) | 12 Months
  Change in walking distance

SECONDARY OUTCOMES:
Technical success of device placement (at exit from procedure room) | Intraprocedural
  * Freedom from mortality
  * Successful access, delivery of the device, and retrieval of the delivery system
  * Correct positioning of the device into the proper anatomical location
  * Freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication
Device success within 30 days after device placement | 1 Month
  * Technical success
  * Freedom from mortality
  * Freedom from surgery or intervention related to the device or to a major vascular or access-related or cardiac structural complication
Procedural success (at 30 days) | 1 Month
  All of the following criteria must be met to be considered a procedural success:
  * Device success (defined above), and
  * Absence of major device or procedure related serious adverse events
Mortality | 12 Months
  Number of days until death
RVAD implantation or heart transplant | 12 Months
  Number of days until Right Ventricular Assist Device (RVAD) implantation or heart transplant
Tricuspid valve surgery or percutaneous tricuspid intervention | 12 Months
  Number of days until tricuspid valve surgery or percutaneous tricuspid intervention
Heart Failure hospitalization or worsening Heart Failure (HF) which encompasses treatment with IV diuretics in the office or Emergency Department treatment during a <24-hour time period | 12 Months
  Number of days until Heart Failure hospitalization or worsening Heart Failure
Kansas City Cardiomyopathy Questionnaire (KCCQ) Score | 12 Months
  Change in KCCQ score (score ranges between 0 and 100)
New York Heart Association (NYHA class) | 12 Months
  Change in NYHA class (range from I to IV)
Six Minute Walking Test (6MWT) | 12 Months
  Change in walking distance

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Kiss, MD, Study Chair — Products & Features GmbH
Locations (36):
- United States (36):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Scripps Memorial Hospital La Jolla, San Diego, California
  - UCSF, San Francisco, California
  - Delray Medical Center, Delray Beach, Florida
  - Largo Medical Center, Largo, Florida
  - Tampa General Hospital, Tampa, Florida
  - Endeavor Health, Glenbrook Hospital, Glenview, Illinois
  - Chicago Advocate Christ, Palos Park, Illinois
  - Ascension Medical Group St. Vincent The Heart Center of Indiana, Indianapolis, Indiana
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Saint Luke's Mid America Heart Institute, Kansas City, Missouri
  - Washington University St Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke Cardiology Clinic, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Oregon Health Services, Portland, Oregon
  - UPMC Pinnacle, Harrisburg, Pennsylvania
  - UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania
  - WellSpan York Hospital, York, Pennsylvania
  - MUSC, Charleston, South Carolina
  - Houston Methodist, Houston, Texas
  - University of Texas (Memorial Hermann), Houston, Texas
  - Intermountain Heart Institute - Intermountain Medical Center, Murray, Utah
  - UVA School of Medicine, Charlottesville, Virginia
  - Sentara Healthcare, Norfolk, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - MedStar Washington Hospital Center, Multiple Locations, Washington
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The dataset generated during and/or analysed during the study will be available upon request from the Clinical Research Organization, Meditrial USA Inc. m.tocchi@meditrial.net Datasets will only be made available through publication, unless disclosure is mandated by law.
Access Criteria: Available on request, Published as a supplement to the results publication.

REFERENCES:
- [Background] Estevez-Loureiro R, Sanchez-Recalde A, Amat-Santos IJ, Cruz-Gonzalez I, Baz JA, Pascual I, Mascherbauer J, Abdul-Jawad Altisent O, Nombela-Franco L, Pan M, Trillo R, Moreno R, Delle Karth G, Salido-Tahoces L, Santos-Martinez S, Nunez JC, Moris C, Goliasch G, Jimenez-Quevedo P, Ojeda S, Cid-Alvarez B, Santiago-Vacas E, Jimenez-Valero S, Serrador A, Martin-Moreiras J, Strouhal A, Hengstenberg C, Zamorano JL, Puri R, Iniguez-Romo A. 6-Month Outcomes of the TricValve System in Patients With Tricuspid Regurgitation: The TRICUS EURO Study. JACC Cardiovasc Interv. 2022 Jul 11;15(13):1366-1377. doi: 10.1016/j.jcin.2022.05.022. Epub 2022 May 17. PMID 35583363
- [Background] Amat-Santos IJ, Estevez-Loureiro R, Sanchez-Recalde A, Cruz-Gonzalez I, Pascual I, Mascherbauer J, Abdul-Jawad Altisent O, Nombela-Franco L, Pan M, Trillo R, Moreno R, Delle Karth G, Blasco-Turrion S, Sanchez-Luna JP, Revilla-Orodoea A, Redondo A, Zamorano JL, Puri R, Iniguez-Romo A, San Roman A. Right heart remodelling after bicaval TricValve implantation in patients with severe tricuspid regurgitation. EuroIntervention. 2023 Aug 7;19(5):e450-e452. doi: 10.4244/EIJ-D-23-00077. No abstract available. PMID 37083622
- [Background] Abdul-Jawad Altisent O, Codina P, Puri R, Bayes-Genis A. Transcatheter bi-caval valve implantation (CAVI) significantly improves cardiac output: mechanistic insights following CardioMEMS(R) and TricValve(R) implantation. Clin Res Cardiol. 2022 Aug;111(8):966-968. doi: 10.1007/s00392-022-02029-8. Epub 2022 May 2. No abstract available. PMID 35499708
- [Result] Chandran K, Long A, Bishop J, Berman P, Matar F, Oliveira GH, Bezerra HG. First In-Man Experience With TricValve Transcatheter Bicaval Valve System in Left Ventricular Assist Device Heartmate II Patient for High-Risk Tricuspid Regurgitation. Circ Heart Fail. 2023 Jun;16(6):e010027. doi: 10.1161/CIRCHEARTFAILURE.122.010027. Epub 2023 Jun 6. No abstract available. PMID 37278243
- See also: Description: Products & Features, manufacturer of TricValve® Transcatheter Bicaval Valve System — https://productsandfeatures.com/
- See also: Meditrial Clinical Research Organization — http://www.meditrial.net